CLINICAL TRIAL: NCT07109193
Title: The Relationship Between Intraperitoneal Drain Placement and Postoperative Pain in Gynecologic Laparoscopy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud qayed mohamed abed, Director, Assiut University
Other Study IDs: Intraperitoneal drain
Record Dates: First submitted 2025-06-26; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Hysterectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the effect of intraperitoneal drain placement on postoperative pain after Gynecologic laparoscopy To evaluate whether the use of drains contributes to improved other clinical outcomes

DETAILED DESCRIPTION:
Operative laparoscopy is becoming the primary approach for treatment of benign gynaecologic diseases, as it is a less invasive procedure and can help shorten the length of hospitalization., Most complications occur during abdominal access or port placement, while other complications arise during abdominal insufflations, tissue dissection, and homeostasis. However, postoperative pain at the shoulder and upper abdomen has been shown to be the most common complaint in many studies. It has been hypothesized that this is due to CO2 residue, which causes stretching of the post distended diaphragm and peritoneum after prolonged surgery. The suprapubic pain comes directly from the surgical wound, which is also affected by postoperative abdominal distension Several methods have been recommended to improve postoperative pain for ambulatory procedures, including a pulmonary recruitment maneuver,intraperitoneal infusions with saline or analgesic drugs,low pressure laparoscopic surgery,and the prescription of different types of preoperative medicine.Studies have shown peritoneal gas drain to be a procedure that could potentially be used to alleviate postoperative pain. Many previous studies have reported good results from using this procedure. Recently, a systematic review mentioned that there was little evidence to support the effectiveness of intraperitoneal gas drain in reducing postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Elective procedure: Patients scheduled for elective pure laparoscopic gynecologic surgery (e.g., ovarian cystectomy, endometriosis resection, diagnostic laparoscopy).
* ASA Physical Status: I-II (i.e., healthy or mild systemic disease).

BMI: 18-35 kg/m².

Informed Consent: Able and willing to give written consent and comply with postoperative pain assessments.

Exclusion Criteria:

1 - Malignancy: Known or suspected gynecologic malignancy requiring staging or radical surgery.

2. Conversion: Intraoperative conversion to laparotomy.

3. Coagulopathy: Bleeding disorders or therapeutic anticoagulation that cannot be paused perioperatively.

4. Prior Major Pelvic Surgery: ≥ 2 previous open abdominal operations (to avoid confounding from adhesions).

5. Intra-Abdominal Infection: Active pelvic inflammatory disease or untreated urinary tract infection.

6. Chronic Pain/Opioid Use: Regular opioid use or chronic pelvic pain syndromes (endometriosis pain > 6 months).

7. Allergy/Contraindication: Allergy to standard analgesics or contraindication to intraperitoneal drain placement (e.g., severe adhesions).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The study population will consist of women undergoing elective laparoscopic gynecologic surgery at [Insert Hospital/Institution Name] over a [insert duration, e.g., 6-month or 12-month] period. Eligible participants will be adult females aged 18 to 65 years who are scheduled for non-oncologic, minimally invasive gynecologic procedures such as ovarian cystectomy, salpingectomy, diagnostic laparoscopy, or laparoscopic management of endometriosis.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Corelation between intraperitoneal drain placement and Postoperative pain in Gynecologic laparoscopy | Baseline
  Evalute post operative pain levels and discomfort through Visual Analouge Scale (VAS) score

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kerimoglu OS, Yilmaz SA, Pekin A, Incesu F, Dogan NU, Ilhan TT, Celik C. Effect of drainage on postoperative pain after laparoscopic ovarian cystectomy. J Obstet Gynaecol. 2015 Apr;35(3):287-9. doi: 10.3109/01443615.2014.948824. Epub 2014 Aug 20. PMID 25140836
- [Background] Abbott J, Hawe J, Srivastava P, Hunter D, Garry R. Intraperitoneal gas drain to reduce pain after laparoscopy: randomized masked trial. Obstet Gynecol. 2001 Jul;98(1):97-100. doi: 10.1016/s0029-7844(01)01383-7. PMID 11430964
- [Background] Swift G, Healey M, Varol N, Maher P, Hill D. A prospective randomised double-blind placebo controlled trial to assess whether gas drains reduce shoulder pain following gynaecological laparoscopy. Aust N Z J Obstet Gynaecol. 2002 Aug;42(3):267-70. doi: 10.1111/j.0004-8666.2002.00267.x. PMID 12230061